CLINICAL TRIAL: NCT00347906
Title: Photodynamic Therapy Versus Transpupillary Thermotherapy in Occult CNV in Age-related Macular Degeneration
Brief Title: Photodynamic Therapy (PDT) Versus Transpupillary Thermotherapy (TTT) in Occult Choroidal Neovascularization (CNV) in Age-related Macular Degeneration (AMD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting patients
Sponsor: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Dnr 00052
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2003-11

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: laser treatment

SUMMARY:
The purpose of this study is to compare the effect of PDT and TTT for the treatment of subfoveal occult CNV in age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* > 55 years of age,
* Subfoveal occult only CNV due to AMD,
* < 4 disc areas or > 4 disc areas
* VA < 0.4

Exclusion Criteria:

* Sign of classic CNV,
* CNV in other diagnoses than AMD,

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Christina I Frennesson, MD, PhD, Principal Investigator — Linkoeping University